CLINICAL TRIAL: NCT05713799
Title: Phase II Trial of the Combination of Alpha-lipoic Acid and Mirabegron in Women and in Men With Obesity
Brief Title: Trial of the Combination of Alpha-Lipoic Acid and Mirabegron in Women and in Men With Obesity
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 10000220; 000220-DK
Record Dates: First submitted 2023-02-03; First posted 2023-02-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11-25

CONDITIONS: Insulin Resistance; Obesity
Keywords: Obesity; Insulin Sensitivity; Insulin Resistance; Placebo
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — mirabegron; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MG+ALA (Active Comparator): Participants take mirabegron + alpha lipoic acid daily for 4 weeks. There is testing pre- and post-treatment. Will evaluate the effects of MG+ALA on metabolic heath.
  Interventions: Drug: Mirabegron; Drug: Alpha-lipoic acid
- MG+Placebo (Placebo Comparator): Participants take mirabegron + placebo daily for 4 weeks. There is testing pre- and post-treatment. Will evaluate the effects of MG+Placebo on metabolic heath.
  Interventions: Drug: Placebo; Drug: Mirabegron

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: MG+Placebo
Drug: Mirabegron — selective beta3-AR agonist approved
Drug: Alpha-lipoic acid — ALA is an antioxidant that is available over the counter
  Arms: MG+ALA

SUMMARY:
Background:

Obesity and related illnesses cause at least 2.8 million deaths each year worldwide. Few treatments exist for obesity that are safe and widely available. A study drug (mirabegron [MG]) combined with a supplement (alpha-lipoic acid [ALA]) may help.

Objective:

To learn how MG and ALA can help the body process food.

Eligibility:

People aged 18 to 65 years with a body mass index between 30 and 40 kg/m2.

Design:

Participants will be screened. They will have a physical exam. They will have blood and urine tests and a test of their heart function. They will speak with a dietician.

The study has two phases. Each phase begins with a 2-day stay in the clinic; then the participant will take the study drugs at home for about 4 weeks, followed by another 2-day stay in the clinic. They will also have outpatient visits about 2 weeks after each clinic stay.

During the clinic stays, participants will undergo many tests:

They will have a plastic tube (catheter) inserted into a vein in each arm. These will be used to draw blood and to infuse glucose (sugar) and insulin.

They will have imaging scans.

They will have a clear hard plastic shield placed over their head to measure oxygen and carbon dioxide as they breathe.

Participants will take the study drugs at home. Both MG and ALA are taken by mouth with water. During one phase, participants will take MG plus a placebo. A placebo looks like the study drug but doesn t contain medicine.

They will log their diet, exercise, and sleep....

DETAILED DESCRIPTION:
Study Description:

This is a single site, Phase II single-blinded, randomized placebo control crossover pilot study. This study aims to explore the effect of adding alphalipoic acid (ALA) to mirabegron (MG) on glucose metabolism and lipolysis rate. MG 50 mg/d with placebo or MG 50 mg/d + ALA will be given to 48 total otherwise healthy women (24) and men (24) with obesity over 4 weeks followed by a 4-12 week washout period, after which subjects cross over to the other treatment. Subjects will undergo metabolic testing, safety assessments, and imaging before and after each of the two treatment cycles. Women and men will be studied separately using the same protocols.

We hypothesize that in women and in men with obesity (BMI 30-40 kg/m2), the increases in insulin sensitivity before and after four weeks of treatment will be higher when subjects are taking the combination MG 50 mg/d and ALA 2.4 g/d compared to when they are taking MG 50 mg/d with placebo. Of note, based on our preliminary data and reports in the literature, a key secondary hypothesis is that in women and in men with Grade 1 and 2 obesity (BMI 30-40 kg/m2), the increases in beta3-AR agonist-induced lipolysis before and after four weeks of treatment will be higher in subjects taking the combination MG 50 mg/d and ALA 2.4 g/d compared to taking MG 50 mg/d + placebo.

Objectives:

Primary objective:

To compare the changes in insulin sensitivity after four weeks of treatment with the combination MG 50 mg/d and ALA 2.4 g/d to the changes after taking MG 50 mg/d + placebo.

Secondary objectives:

* Assess the rate of steady-state whole-body lipolysis measured as the rate of isotope appearance (Ra) of [2H5] glycerol before and on treatment compared to MG + placebo. While not optional, these studies are dependent on the availability of [2H5] glycerol.
* Determine serum lipids levels before and on treatment compared to MG + placebo
* To determine the safety and tolerability of the combination of ALA at dose 2.4 g/d given with mirabegron (MG, 50 mg/d).
* Assess adipose tissue inflammation and serum inflammatory markers before and on treatment compared to MG + placebo

Exploratory Objectives (optional):

* Assess the resting metabolic rate (RMR) before and on treatment compared to MG + placebo
* Assess body composition before and on treatment compared to MG + placebo
* Assess changes in glucose turnover using labeled glucose and water before and on treatment compared to MG + placebo
* Assess liver inflammation and fat content by MRS/MRE before and on treatment compared to MG + placebo

Endpoints:

Primary Endpoint: the changes in the Insulin Sensitivity Index (SI) obtained from the FSIGT.

Secondary Endpoints:

* Maximum observed plasma concentration of ALA (Cmax), time to maximum observed plasma concentration of ALA (Tmax), and area under the
* concentration-time curve from 0 to 6 hours post-dose.
* The number of subjects that develop Serious or non-serious AEs during and 2 weeks after treatment.
* Changes in adipose tissue local inflammation (crown-like structures) before and on treatment will be compared between the two study arms.
* Changes in serum cytokines (IL-6, TNFalpha, IL-17A, IL-10), CRP before and after treatment will be compared between the two study arms.
* Changes in plasma lipids before and after treatment will be compared between the two study arms.
* The rate of steady-state whole-body lipolysis measured as the rate of isotope appearance (Ra) of [2H5] glycerol before and on treatment will be compared between the two study arms.

Exploratory endpoints

* Anterior abdominal wall adipose tissue-resident immune cells
* Liver inflammation and fibrosis via MR
* Bone marrow adipose tissue BMAT via MR
* Resting metabolic rate (RMR). respiratory quotient (RQ), % body fat
* Gluconeogenesis and glucose turnover using stable isotopes

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Adult subjects aged 18 - 65 years
2. BMI greater than 30 kg/m2 and less than 40 kg/m2

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Type 1 diabetes mellitus; type 2 diabetes mellitus; or any person taking exogenous insulin therapy or any medication that increases risk of hypoglycemia
2. Pregnancy, childbirth within the last year, or breastfeeding in the past 12 months (for women only)
3. Hemoglobin <= 10 g/dl, Platelets <= 75 x 10^9 per liter, white blood cell count <= 4 x 10^9 per liter) or patients with eGFR <60 ml/min/1.72 m2 and a Urine Albumin Creatinine Ratio >300 mg/g
4. Since recent weight loss would change the metabolic rate, subjects that have been on a very low-calorie diet (<800 kcal/d) within a year or self-reported weight loss >5% in the preceding six months.
5. Trained athletes
6. History of seizure disorder
7. An active history of abnormal bladder function, diagnosis of bladder outlet obstruction, urgency, and urinary frequency or use of antimuscarinic medication to treat overactive bladder (OAB)
8. History of hypertension or subjects on antihypertensive therapy since the combination therapy on other beta receptors is unknown.
9. Medication that causes QT prolongation, adrenergic agonists, cardiac beta-blockers, calcium channel blockers, insulin resistance (systemic corticosteroids), monoamine oxidase, or medications known to be CYP2D6 substrates
10. Current use of medications/dietary supplements/alternative therapies known to alter energy metabolism, including levothyroxine.
11. Subjects with moderate hepatic impairment (Child-Pugh Class B) or above
12. Unable to take oral medication
13. Individuals with significant medical comorbidities that would render the subject s participation unsafe as assessed by the investigator
14. Individuals with cardiac arrhythmia or abnormal baseline EKG
15. Individuals who have current substance abuse or a psychiatric disorder or any other condition that, in the investigators' opinion, would impede competence, compliance, or participation in the study.
16. Individuals with known allergies to mirabegron and alpha-lipoic acid or sulfa containing drugs
17. Inability to provide informed consent
18. Other factors that the PI will determine to affect the safety or outcome of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
changes in the Insulin sensitivity index (SI) obtained from FSIGT | 4 weeks after intervention
  changes in the Insulin sensitivity index

SECONDARY OUTCOMES:
Maximum observed plasma concentration of ALA (Cmax), time to maximum observed plasma concentration of ALA (Tmax), and area under the concentration-time curve. | 4 weeks after intervention
  Maximum observed plasma concentration of ALA

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Cypess, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000220-DK.html